CLINICAL TRIAL: NCT03961230
Title: Oral Chinese Herbal Medicine for Psoriasis Vulgaris With Blood Heat Syndrome: a Randomised, Double-blind, Doubledummy, Multicentre Clinical Trial
Brief Title: Oral Chinese Herbal Medicine for Psoriasis Vulgaris With Blood Heat Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Collaborators: Beijing Hospital of Traditional Chinese Medicine (Other); First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Unknown); Gansu University of Chinese Medicine (Other); Guangxi Zhuang Autonomous Region Dermatology Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018YFC1705302
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Psoriasis Vulgaris
Keywords: Psoriasis Vulgaris; Jueyin granules; Blood heat syndrome; Randomized controlled trial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Chinese medicine (Experimental): Participants in experimental group will receive Jueyin granule two times daily after meals three times per week for 8 weeks.
  Interventions: Drug: Jueyin granules
- Oral Chinese medicine placebo (Placebo Comparator): Participants in placebo group will receive Jueyin granule placebo two times daily after meals three times per week for 8 weeks.
  Interventions: Drug: Jueyin Granules Placebo

INTERVENTIONS:
Drug: Jueyin granules — Put each bag of medicine in the same amount into the same container, pour about 50 ml of warm water, stir until the particles are basically dissolved, and then add appropriate amount of boiling water to dilute.
  Other Names: Chinese Herbal Medicine
  Arms: Oral Chinese medicine
Drug: Jueyin Granules Placebo — Put each bag of medicine in the same amount into the same container, pour about 50 ml of warm water, stir until the particles are basically dissolved, and then add appropriate amount of boiling water to dilute.
  Other Names: Chinese Herbal Medicine
  Arms: Oral Chinese medicine placebo

SUMMARY:
We designed this study as a multicenter, randomized, double blinded and placebo-controlled clinical trial. The aim of the study is to evaluate the clinical efficacy, safety and control of recurrence rate of psoriasis with blood stasis syndrome.

DETAILED DESCRIPTION:
Psoriasis is a chronic, relapsing, inflammatory, multisystem disease characterized by infiltration of inflammatory cells, hyperplasia of epidermal keratinocytes, and abnormal differentiation. Latest data estimate that the prevalence of psoriasis in adults has increased to 11.43%, which shows that the control and treatment of psoriasis is still insufficient. Recent studies showed that traditional Chinese medicine (TCM) is one of the effective methods for the treatment of psoriasis. More and more evidences support the recognition of psoriasis not only affects the skin, but also suffers a chronic multisystem inflammation. Chinese medicine believes that the blood heat is the root of the onset of psoriasis, so the treatment of psoriasis should focus on the method of clearing heat and cooling blood. Therefore, the method of promoting clearing heat and cooling blood. has always been the focus of TCM treatment and prevention of psoriasis. This multicenter, randomized, double-blind, placebo-controlled trial will provide high-quality clinical evidences for evaluating the efficacy, safety and recurrence rate of Jueyin granule, a representative prescription for the treatment of psoriasis with blood heat syndrome, in the treatment of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Comply with the diagnostic criteria of Western medicine for psoriasis and the diagnostic criteria for TCM syndromes;
2. Skin lesions involve ≤10% BSA (the lesions are mainly located in the trunk and/or limbs, palm/sole, face/scalp, vulva area is not included);
3. Age between 18 and 65 years old;
4. Those who voluntarily participate in the study and sign informed consent.

Exclusion Criteria:

1. Patients with erythrodermic, arthritic, pustular or punctate psoriasis;
2. Other active skin diseases may affect the condition assessment;
3. Received research drugs, biological agents and immunosuppressive agents within 1 month;
4. 2 weeks of treatment with topical glucocorticoids, phototherapy, etc.;
5. During severe, uncontrollable local or systemic acute or chronic infections;
6. Patients with severe systemic diseases; or clinical test indicators in one of the following conditions: alanine aminotransferase or aspartate aminotransferase increased by >1.5 times the upper limit of normal; creatinine increased by 1.5 times the upper limit of normal; blood routine indicators (white blood cell count) Any one of the red blood cell count, hemoglobin amount, and platelet count) is below the lower limit of normal; or other laboratory abnormalities are judged by the investigator to be unsuitable for participation in the trial;
7. A history of malignant tumors and patients with primary or secondary immunodeficiency and hypersensitivity;
8. Such surgery will be required during major surgery or study during 8 weeks;
9. Pregnant or lactating women;
10. A person with a history of alcohol abuse, drug abuse or drug abuse;
11. Have a history of serious mental illness or family history;
12. Other reasons researchers believe that it is inappropriate to participate in this research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Psoriasis area and severity index | Up to 56 days after treatment.
  Psoriasis Area and Severity Index involves grading psoriatic plaques based on erythema (E), infiltration (I), desquamation (D). Severity is graded from 0-4 for each criteria (0 - none, 1 - slight, 2 - moderate, 3 - severe, and 4 - very severe). The body is divided into 4 regions, head, upper extremities, trunk, and lower extremities, and for each region, the surface area involvement is graded on a 0-6 scale (0 - 0% involvement, 1 - <10%, 2 - 10-<30%, 3 - 30-<50%, 4 - 50-<70%, 5 - 70-<90%, 6 - 90-100%).The highest potential PASI score is 72, with higher PASI scores indicating worse psoriasis.

SECONDARY OUTCOMES:
Body surface area (BSA) | Up to 56 days after treatment.
  The percentage of BSA involved in psoriasis is estimated by fingerprinting, where the entire palm of the patient represents approximately 1% of the total BSA. The number of handprints on psoriasis skin in a body part is used to determine the extent to which the body part is affected by psoriasis (%)
Physician Global Assessment (PGA) | Up to 56 days after treatment.
  Physician Global Assessment (PGA) is scored on a 5-point scale, reflecting a global consideration of the erythema (E), infiltration (I), desquamation (D) across all psoriatic lesions. It is calculated as follows: PGA score = (E + I + D) / 3, then the score needs to be rounded to the nearest whole number [PGA scale: Clear (0) - Very Severe (5)].
Dermatology Life quality index(DLQI) | Up to 56 days after treatment.
  The Dermatology Life Quality Index (DLQI) is a participant-reported questionnaire used to measure the health-related quality of life (QOL) of adults suffering from a skin disease. Scores range from 0-30, a higher score indicating a greater impact on a participant's quality of life.
Patient-reported quality of life (PRQoL) | Up to 56 days after treatment.
  PRQoL is used to assess the impact of psoriasis on individual social life. Scores range from 0-25, a higher score indicating a greater impact on a participant's social life.
Visual Analogue Score (VAS) | Up to 56 days after treatment.
  Visual Analog Scale (VAS) is used to measure lesion pruritus from 0 to 100 mm at eash visit (with 0 being no pruritis and 100 being maximum pruritis).
TCM symptom score | Up to 56 days after treatment.
  The TCM symptom score is used to assess changes in blood syndrome related symptoms during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Zhou, Study Chair — Department of dermatology, Shanghai Yueyang Integrated Medicine Hospital, Shanghai
Locations (4):
- China (4):
  - First Affiliated Hospital of Anhui University of Traditional Chinese Medicine, Hefei, Anhui
  - Beijing Hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Affiliated Hospital of Gansu University of Chinese Medicine, Nanchang, Gansu
  - Guangxi Zhuang Autonomous Region Dermatology Hospital, Nanning, Guizhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li S, Zhang C, Zhang HY, Zhou M, Wang SN, Xu R, Zhou DM, Ji YR, Lv JJ, Yin QF, Wang RP, Li W, Liu YP, Wang JF, Li B, Li X. Efficacy and Safety of Jueyin Granules for Patients with Mild-to-Moderate Psoriasis Vulgaris: Protocol for a Multicenter Randomized Placebo-Controlled Trial. Evid Based Complement Alternat Med. 2020 Apr 9;2020:8942301. doi: 10.1155/2020/8942301. eCollection 2020. PMID 32351609